CLINICAL TRIAL: NCT03425799
Title: Efficacy and Safety of Tranexamic Acid in Spinal Fusion Surgery
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Low recruitment rate
Sponsor: Exela Pharma Sciences, LLC. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CP-006-2017
Record Dates: First submitted 2018-01-23; First posted 2018-02-08 (Actual); Results first posted 2021-06-21 (Actual); Last update posted 2021-06-21 (Actual); Status verified 2020-09

CONDITIONS: Spinal Fusion
MeSH Terms: interventions — Sodium Chloride; Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Sodium Chloride 0.9% (Placebo Comparator): Sodium Chloride 0.9% infused at 3 mL/kg over one hour followed by continuous infusion at 0.3 mL/kg for maximum infusion volume of 5 mL/kg
  Interventions: Drug: Sodium Chloride 0.9% Inj
- Tranexamic Acid 10 mg/mL (Experimental): Tranexamic Acid 10 mg/mL infused at 3 mL/kg over one hour followed by continuous infusion at 0.3 mL/kg for maximum infusion volume of 5 mL/kg
  Interventions: Drug: Tranexamic Acid

INTERVENTIONS:
Drug: Sodium Chloride 0.9% Inj — Inactive ingredient mixture for injection without drug, intravenous infusion bags containing normal saline, manufactured and provided by Exela Pharma Sciences, LLC from a single batch / lot.
  Other Names: Saline
  Arms: Sodium Chloride 0.9%
Drug: Tranexamic Acid — Tranexamic Acid Intravenous Infusion Bags (10 mg/mL), manufactured and provided by Exela Pharma Sciences, LLC from a single batch / lot.
  Other Names: Tranexamic Acid in 0.7% sodium chloride
  Arms: Tranexamic Acid 10 mg/mL

SUMMARY:
The purpose of this study is to see if Tranexamic Acid can safely reduce bleeding in people undergoing spinal fusion surgery.

DETAILED DESCRIPTION:
This will be a multicenter, randomized, double-blind, parallel group study comparing tranexamic acid (test) to placebo (control) for reduction of perioperative blood loss after complex spinal fusion surgery (defined as T2 to Pelvis/Sacrum and greater than 4 Functional Spinal Units (4 discs/motion segments=5 Vertebral segments)). In addition to test and control treatments, all patients undergoing spinal fusion surgery will receive anesthesia and standard of care for blood loss including colloid/crystalloid fluid replacement and packed red cells, if necessary, according to a common multi-institutional protocol. Anesthesia will keep the mean arterial pressure as low as safe for the patient during exposure of surgery (estimated at 60-80 MAP). Patients will be randomized to receive either 30 mg/kg tranexamic acid as a one hour infusion (3 mL/kg) loading dose prior to start of procedure and as an infusion at 3 mg/kg/h (0.3 mL/kg/h) of tranexamic acid throughout the surgery in the test group; or, a one hour infusion at 3 mL/kg of 0.9% saline prior to start of the procedure and an infusion of 0.9% saline at 0.3 mL/kg/h in the control group. The maximum total dose will be 50 mg/kg.

The active phase of the study will be until discharge postoperatively for efficacy measurements and at 6 weeks for safety follow-up. The randomization will be open only to the statistician generating the randomization sequence. All PI(s), study conduct and monitoring staff, as well as the subjects will be completely blinded to the treatments except in the case of emergency.

The study will be terminated if ≥5/12 or 10/36 patients enrolled in the study are diagnosed with treatment related serious adverse events.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients (Male or Female) over age eighteen (>18) electively undergoing complex spinal fusion surgery (defined as T2 to Pelvis/Sacrum and greater than 4 Functional Spinal Units (4 discs/motion segments=5 Vertebral segments).
* Female subjects of childbearing potential with a negative serum (beta human chorionic gonadotropin [HCG]) pregnancy test at screening and urine pregnancy test at each admission; who are not breastfeeding; do not plan to become pregnant during the course of the study; and agree to use an approved method of birth control, such as condoms, foams, jellies, diaphragm, intrauterine device, sexual abstinence for at least 3 months prior to study
* Able to provide written informed consent after risks and benefits of the study have been explained
* Able to communicate effectively with study personnel.

Exclusion Criteria:

* History or presence of any clinically significant (based on the Investigator's judgment) cardiovascular, respiratory, metabolic, hepatic, gastrointestinal, renal, hematological, dermatological, neurological, or psychiatric disease or condition preventing the use of tranexamic acid
* History of renal failure or elevated creatinine above 1.4
* Any diagnosis of spinal tumor or intradural pathology
* Diagnosis of ankylosing spondylitis
* History or presence of acquired disturbance of color vision
* History of seizures
* History of thromboembolic event (DVT or PE) within the past year
* Current use of anticoagulant medications or past medical history leading to an abnormal coagulation profile preoperatively
* Subjects diagnosed with fibrinolytic disorders requiring intra-operative antifibrinolytic treatment; hematological disease (thromboembolic events, hemoglobinopathy, coagulopathy, or hemolytic disease)
* Significant drug sensitivity or significant allergic reaction to any drug, including tranexamic acid, based on the Investigator's judgment
* A subject who has donated or lost 450 mL or more blood volume (including plasmaphoresis) or had a transfusion of any product within 3 months prior to the initial study drug administration
* Pre-operative anemia (hb <110 in females, Hb <120 in males)
* Any subject that chooses to refuse blood products for ethical or religious purposes (Jehovah's Witness)
* Current participation in a drug or other investigational research study or participation within 30 days prior to the initial study drug administration
* A subject who may not be able to comply with the safety monitoring requirements of this clinical trial or is considered by the investigator, for any reason, to be an unsuitable candidate for the study.
* Intraoperative cardiovascular, pulmonary, orthopedic, or anesthetic complication such as myocardial infarction, intraoperative fracture, vasopressor support or emergent intubation.
* Female patients who are using combination hormonal contraception.
* Patients with history of subarachnoid hemorrhage.
* Patients with serum creatinine above upper limit of normal (ULN).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2018-10-17 (Actual); Primary Completion 2019-10-23 (Actual); Study Completion 2020-01-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neel Anand, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (4):
- United States (4):
  - Memorial Orthopaedic Surgery Group, Long Beach, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Rush University Medical Center - Division of Spine Surgery, Chicago, Illinois
  - Spine Care Orthopedics - NYU Lagone Medical Center, New York, New York

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study terminated due to low recruitment
Pre-assignment Details: Study terminated due to low recruitment
Groups:
- Placebo: Placebo (0.9% Sodium Chloride) infused at 3 mL/kg over one hour followed by continuous infusion at 0.3 mL/kg for maximum infusion volume of 5 mL/kg
  Placebo Intravenous Infusion Bags, manufactured and provided by Exela Pharma Sciences, LLC from a single batch / lot.
Period: Overall Study
Arm/Group | Tranexamic Acid 10 mg/mL | Placebo
Started | 0 (Study terminated due to low recruitment) | 0 (Study terminated due to low recruitment)
Completed (Study terminated due to low recruitment) | 0 (Study terminated due to low recruitment) | 0 (Study terminated due to low recruitment)
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Not Available. Study Terminated and data were not collected.
Groups:
- Total: Total of all reporting groups
Arm/Group | Sodium Chloride 0.9% | Tranexamic Acid 10 mg/mL | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Continuous
Sex: Female, Male
Race (NIH/OMB)
Total Blood Loss

OUTCOME MEASURES:

1. Primary Outcome: Total Blood Loss
Description: The Total Blood Loss will be estimated based on the hemoglobin content of the blood prior to surgery (mg/dL) and at each of the desired post-surgery time-points (mg/dL). Blood samples for hemoglobin measurement will be collected prior to start of procedure, at the end of the procedure, at 24 h, and every 24 h thereafter until discharge and removal two subfascial drains.
Time Frame: From time of surgery until discharge
Population: Data were not collected
Arm/Group | Sodium Chloride 0.9% | Tranexamic Acid 10 mg/mL
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Incidence of Autologous or Allogenic Blood Transfusion
Description: Number of Units of autologous transfusion and allogenic transfusion
Time Frame: From time of surgery until discharge
Population: Study was terminated due to low recruitment. Data were not collected.
Arm/Group | Sodium Chloride 0.9% | Tranexamic Acid 10 mg/mL
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Total Measured Blood Loss
Description: Estimated as 3x cell saver
Time Frame: From time of surgery up to 24 hours after surgery
Population: Total number of patients recruited and treated was 5 patients. No analyses were performed due to early termination of the study due to low recruitment.
Arm/Group | Sodium Chloride 0.9% | Tranexamic Acid 10 mg/mL
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Number of Patients With Symptomatic Anemia Precipitated Transfusion
Description: Number of patients with symptomatic anemia precipitated transfusion in each group
Time Frame: Until discharge
Population: as for outcome 3
Arm/Group | Sodium Chloride 0.9% | Tranexamic Acid 10 mg/mL
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Number of Patients With Adverse Events Related to Tranexamic Acid
Description: Number of patients with adverse events related to tranexamic acid in each group
Time Frame: up to 6 weeks
Population: as for outcome 3
Arm/Group | Sodium Chloride 0.9% | Tranexamic Acid 10 mg/mL
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Data not collected
Description: Data not collected
Arm/Group | Sodium Chloride 0.9% | Tranexamic Acid 10 mg/mL
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-29): https://cdn.clinicaltrials.gov/large-docs/99/NCT03425799/Prot_SAP_001.pdf